CLINICAL TRIAL: NCT07398794
Title: Evaluation of Combining Video Feedback Teaching With Virtual Simulation for Ceramic Veneer Tooth Preparation: A Prospective Randomized Controlled Study
Brief Title: Video Feedback Teaching With Virtual Simulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jiangsu Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: JiangsuMC
Record Dates: First submitted 2026-01-27; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Ceramic Veneer; Head Simulator; Video Feedback Teaching; Virtual Simulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Teaching (Active Comparator): This group received the traditional teaching method. This included theoretical instruction, a live clinical demonstration by an instructor, followed by guided and independent hands-on practice sessions on head simulators.
  Interventions: Behavioral: Traditional Teaching Method
- Video Feedback with Virtual Simulation (Experimental): This group received the video feedback teaching method combined with virtual simulation. After theoretical instruction, they completed a virtual simulation module. The instructor's live demonstration was recorded. Students then practiced in pairs, recorded each other, and reviewed the videos for peer and instructor critique.
  Interventions: Behavioral: Video Feedback Teaching combined with Virtual Simulation

INTERVENTIONS:
Behavioral: Traditional Teaching Method — The intervention consisted of a 20-minute theoretical instruction on ceramic veneer preparation, followed by a 20-minute live clinical demonstration by an instructor. Students then engaged in supervised and independent hands-on practice sessions (100 minutes each on two consecutive days) using head simulators, during which the instructor provided immediate feedback.
  Arms: Traditional Teaching
Behavioral: Video Feedback Teaching combined with Virtual Simulation — The intervention included a 20-minute theoretical instruction and completion of a mandatory virtual simulation module. After a live instructor demonstration (recorded on video), students practiced in pairs, recording each other's procedures. They then conducted peer critiques by reviewing the videos. An instructor-led group video review session provided further feedback. A second day involved additional practice with instructor guidance.
  Arms: Video Feedback with Virtual Simulation

SUMMARY:
This study aims to evaluate the effectiveness of a combined teaching method using video feedback and virtual simulation for training dental students in ceramic veneer tooth preparation, compared to traditional teaching methods. The hypothesis is that this integrated approach will lead to better acquisition of practical skills.

The study is designed as a prospective, randomized controlled trial. Forty dental students about to begin their clinical internship will be randomly assigned to one of two groups. One group will receive traditional teaching involving lectures and instructor-led demonstrations on dental simulators. The other group will receive the experimental intervention, which combines the use of a virtual simulation training module with video recording of hands-on practice sessions. In the experimental group, students will review their recorded performances for self and peer assessment under instructor guidance.

All participants' ceramic veneer preparation skills will be assessed before the training begins. Their skills will then be re-evaluated at 1 month, 2 months, and 3 months after completing the training. The assessments will focus on two main areas: the ergonomic quality of the student's operating posture and the technical quality of the tooth preparation they perform on a simulator.

ELIGIBILITY:
Inclusion Criteria:

* Prospective dental students from Jiangsu Medical College who were about to start clinical internships.
* Students who have completed theoretical and practical coursework in the dental profession.
* Students who are about to undergo pre-service training for clinical placements.

Exclusion Criteria:

* Not applicable

Ages: 17 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Tooth Preparation Morphology Score | Assessed at baseline (before training), and at 1 month, 2 months, and 3 months after the start of training.
  Score assessing the quality of the ceramic veneer tooth preparation. Based on five criteria: amount of tooth preparation (neck and shoulder preparation), positioning of the neck and shoulder, smoothness and continuity of the shoulder, finishing and polishing of the preparation, and damage to the gum or adjacent teeth. Each criterion is scored out of 20 points, with a total possible score of 100. Higher scores indicate better quality.
Operating Position Score | Assessed at baseline (before training), and at 1 month, 2 months, and 3 months after the start of training.
  Score evaluating ergonomic posture during the preparation procedure using the Modified Dental Operator Posture Assessment Instrument (M-DOPAI). It includes 12 scoring items related to six body parts (back, hands, shoulders, neck, head, and feet). Scores range from 12 to 32, with lower scores indicating better posture.

SECONDARY OUTCOMES:
Student Feedback Questionnaire Score | Administered after the completion of the training period (after the 3-month assessment).
  A questionnaire administered to students in the study group to evaluate their perception of the combined video feedback and virtual simulation teaching method. It consists of six statements (e.g., enhanced teacher-student communication, increased interest) rated on a 5-point Likert scale (1=completely disagree, 5=completely agree). Higher scores indicate more positive feedback.

CONTACTS AND LOCATIONS:
Overall Officials: Hao Yu, Master's degree, Principal Investigator — Jiangsu Medical College
Locations (1):
- Hao Yu, Yancheng, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No